CLINICAL TRIAL: NCT00001876
Title: Pulmonary Fibrosis Associated With Rheumatoid Arthritis: Definition of the Natural History of Disease
Brief Title: Lung Disease Associated With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990056; 99-HG-0056
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Fibrosis
Keywords: Interstitial Lung Disease; Collagen Vascular Disease; Extracellular Matrix; Pulmonary Function; DTPA Lung Clearance Scan; Natural History
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases, Interstitial; Collagen Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Combo: Patients with rheumatoid arthritis and biopsy-proven pulmonary fibrosis.
- pulmonary fibrosis: Patients with biobsy-proven idiopathic pulmonary fibrosis only.
- rheumatoid arthritis: Patients with rheumatoid arthritis only.

SUMMARY:
Pulmonary fibrosis (PF) is a condition in which the lungs of a patient become scarred and fibrous. It has been known to occur in as many as 40% of patients diagnosed with rheumatoid arthritis (RA). The cause of the pulmonary fibrosis in patients with RA is unknown.

Patients participating in this study will undergo a series of tests and examinations before and throughout the study. The tests include blood and urine tests, electrical measures of heart function (ECG), chest x-rays, CAT scans, nuclear medicine scans, breathing tests, exercise tests, and fiberoptic bronchoscopy.

The goals of this study are to:

1. Estimate how common pulmonary fibrosis is in patients with rheumatoid arthritis,
2. Describe the natural course of pulmonary fibrosis in patients with rheumatoid arthritis,
3. Estimate the survival rate of patients with pulmonary fibrosis and rheumatoid arthritis, and
4. Learn more about the factors that contribute to the development or progression fibrotic lung disease....

DETAILED DESCRIPTION:
Pulmonary fibrosis is an extra-articular manifestation of rheumatoid arthritis whose etiology remains uncertain. Although the clinical course of many individuals with this disorder can mimic that observed in patients with idiopathic pulmonary fibrosis, the natural history of fibrotic lung disease associated with rheumatoid arthritis remains largely undefined. It is the intent of this clinical protocol to (1) estimate the prevalence of pulmonary fibrosis in individuals with rheumatoid arthritis, (2) define the natural history of pulmonary fibrosis in patients with rheumatoid arthritis, (3) estimate the survival rate of individuals with pulmonary fibrosis and rheumatoid arthritis, and (4) examine pulmonary physiologic, radiologic, and biochemical markers that predict the development or progression of fibrotic lung disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Non-smokers (never smoked or no smoking within the previous 2 years) who are 21 years of age or older with any of the following:

Rheumatoid arthritis with biopsy-proven pulmonary fibrosis or;

Rheumatoid arthritis only, or;

Biopsy-proven idiopathic pulmonary fibrosis.

EXCLUSION CRITERIA:

Forced expiratory volume in one second (FEV1) less than 1L.

Inhalational exposure to fibrogenic fibers or dusts (e.g., asbestos, silica, coal, beryllium).

Chronic cardiopulmonary disorders other than pulmonary fibrosis.

Other collagen vascular disorders (e.g., systemic lupus erythematosus, scleroderma, polymyositis, mixed connective tissue disease).

Non-rheumatoid arthritis.

Viral infections associated with pulmonary fibrosis (e.g., hepatitis B, hepatitis C, human immunodeficiency virus).

Uncorrectable bleeding diathesis.

Pregnancy or lactation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will include individuals with (1) rheumatoid arthritis and biopsy-proven pulmonary fibrosis, (2) rheumatoid arthritis-only, and (3) biopsy-proven idiopathic pulmonary fibrosis-only.@@@
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 1999-04-05 (Actual); Primary Completion 2005-11-09 (Actual); Study Completion 2007-12-11 (Actual)

PRIMARY OUTCOMES:
Prevalence | Ongoing
  To estimate the prevalence of pulmonary fibrosis in individuals with rheumatoid arthritis. Subjects will include patients that have rheumatoid arthritis-only.
Natural History | Ongoing
  To define the natural history of pulmonary fibrosis associated with rheumatoid arthritis in a prospective, longitudinal study.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette R Gochuico, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1999-HG-0056.html